CLINICAL TRIAL: NCT06354192
Title: Data-driven Personalization for Inclusive Outreach and Equitable Outcomes in a Digital Health Intervention for Hypertension Management: A Prospective Observational Study
Brief Title: Precision Nudging for Hypertension Management: Observational Study
Status: Recruiting | Type: Observational
Sponsor: Lirio (Industry)
Collaborators: Cone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 0450
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: Medication adherence; Self-monitoring of blood pressure; Clinical encounters; Health equity; Precision nudging; Digital health intervention; Behavioral reinforcement learning
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Precision Nudging for Hypertension Management: All participants in this study will receive the digital health intervention.
  Interventions: Behavioral: Precision Nudging for Hypertension Management

INTERVENTIONS:
Behavioral: Precision Nudging for Hypertension Management — The hypertension digital health intervention under study combines behavioral science theory with a type of machine learning called reinforcement learning to enable precision nudging: the selection, assembly, and delivery of behavioral science-based messages created to address barriers to, and promote, management of hypertension. The behavioral design process used for the hypertension DHI intentionally includes research on traditionally underserved populations, such as racial and ethnic minorities and people with lower incomes or educational attainment. By including the right ingredients to meet a diverse set of needs and by effectively personalizing the content each individual sees based on their own reactions, the intervention aims to improve health equity by matching each individual to the right behavioral approach.
  Other Names: Digital Health Intervention; Artificial Intelligence Driven Intervention

SUMMARY:
The purpose of the proposed observational study is to explore the relations between data-driven personalization and equitable health outcomes in a digital health intervention (DHI) for hypertension management. In the current intervention, behavioral reinforcement learning is applied to personalize intervention content to maximize the behavioral outcomes of three target behaviors critical for effective hypertension management: clinical encounters, medication adherence, and self-monitoring of blood pressure (SMBP).

ELIGIBILITY:
Inclusion Criteria:

* Patient of Cone Health.
* Hypertension condition considered "uncontrolled" (signaled by an eligibility indicator).
* Most recent blood pressure reading is at or higher than 160/90 (lowered to 140/90 in April 2025 in accordance with approved protocol)

Exclusion Criteria:

* Non-English speaking.
* Globally unsubscribed.
* Locally unsubscribed.
* Deceased.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study will follow participants enrolled in a digital health intervention for hypertension management at one of nine Cone Health Community Access Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical encounter behavioral outcome | 0-18 months
  Adherence with recommended clinical encounters given eligibility based on blood pressure readings and medication
Blood pressure reading clinical outcome | 0-18 months
  Blood pressure reading

SECONDARY OUTCOMES:
Engagement | 0-18 months
  Digital engagement (opens, clicks, responses, etc.)
Medication adherence behavioral outcome | 0-18 months
  Self-reported medication adherence
Self-monitoring of blood pressure behavioral outcome | 0-18 months
  Self-reported self-monitoring of blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Cone Health clinics, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.